CLINICAL TRIAL: NCT01591187
Title: The Feasibility of Text Messaging to Assess Secondhand Smoke Exposure Among Youngsters With Cancer or Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: San Diego State University (Other); University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: XPD12-026 SMTEXT
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Cancer; Sickle Cell Disease
Keywords: Text messaging; Secondhand smoke exposure
MeSH Terms: conditions — Neoplasms; Anemia, Sickle Cell | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cancer: Participants with a diagnosis of cancer.
- Sickle Cell Disease: Participants with a diagnosis of sickle cell disease.
  Interventions: Text messaging, Questionnaire, Interviews
  Interventions: Other: Text messaging; Other: Questionnaire; Other: Interviews

INTERVENTIONS:
Other: Text messaging — Participants report on the smoking that takes place in their presence for a period of 7 days by responding to daily texted messages sent by the research team to their mobile phones. Parents will also be asked to report on the child's SHSe during the same 7-day period so that child and parent reports can be compared.
  Groups: Sickle Cell Disease
Other: Questionnaire — Child and parent questionnaire data about attitudes, behavioral practices to control SHSe, and other socio-environmental factors will be obtained.
  Groups: Sickle Cell Disease
Other: Interviews — Individual interviews with youngsters will provide additional qualitative information about the social context and conditions in the child's environment that maintain or contribute to avoidance of exposure.
  Groups: Sickle Cell Disease

SUMMARY:
Exposure to secondhand smoke is a leading preventable cause of child morbidity and mortality, and the adverse health consequences of secondhand smoke are magnified among youngsters with cancer and sickle cell disease. Current methods for measuring secondhand smoke exposure (SHSe) rely on retrospective reports over extended time periods that are subject to recall errors and systematic inaccuracies in reporting and often do not include the youngster as the primary informant. These methods may underestimate the extent of cumulative SHSe and are not well suited to capturing exposure over time and across settings where young people frequent. More appealing methods that engage youngsters to better monitor tobacco smoke in their environment are warranted.

The study will examine the feasibility of cell phone texting to obtain measures of secondhand smoke exposure (SHSe) in children treated for cancer or sickle cell disease (SCD).

DETAILED DESCRIPTION:
Children participating on this study will be asked to report on the smoking that takes place in their presence for a period of 7 days by responding to daily texted messages sent by the research team to their mobile phones. Rates of participation on the study, compliance with reporting SHSe, and feedback about the technical viability and satisfaction with the texting methods will be obtained. Parents will also be asked to report on the child's SHSe during the same 7-day period so that child and parent reports can be compared. In addition to quantitative child and parent reports of SHSe, child and parent questionnaire data about attitudes, behavioral practices to control SHSe, and other socio-environmental factors will be obtained. Individual interviews with youngsters will provide additional qualitative information about the social context and conditions in the child's environment that maintain or contribute to avoidance of exposure. This information will be collectively used to develop a larger trial that will test a behavioral intervention to reduce SHSe among youngsters with cancer and SCD and require them to monitor their SHSe using text messaging. Measuring SHSe in these vulnerable populations and intervening to reduce their SHSe is critical to protecting their current and long-term health.

As participation rates and compliance may differ among youngsters diagnosed with cancer and sickle cell disease, participants will be stratified by disease group (up to 55 with cancer and up to 55 with SCD).

ELIGIBILITY:
Inclusion Criteria:

* Child Participant:

  * St. Jude Children's Research Hospital (SJCRH) patient with primary diagnosis of any type of cancer or any sickle cell disease genotype (HbSS, HbSC, HbSβ°thal, HbSβ+thal, HbSD, HbSO, Hb S/HPFH, HbSE).
  * 10 to < 18 years of age at the time of enrollment.
  * For cancer patients, at least one month from diagnosis and in active treatment section at the time of enrollment.
  * Lives in a smoking household defined as at least one adult (> 18 years) smoker who resides in the home. Smoking adults will be defined as those who have smoked at least one cigarette in the past 30 days, per parent report.
  * Does not currently use tobacco (defined as abstinence from tobacco during the 30 days preceding the screening assessment as based on patient and/or parent report).
  * Able to demonstrate satisfactory texting skills via mobile phone as determined by study research staff.
  * Cannot have significant cognitive or learning impairment that precludes completion of study measures.
  * Reads and speaks English.
  * Willing and able to provide assent according to institutional guidelines.
* Parent Participant:

  * Parent of SJCRH patient who meets criteria as stated above.
  * Reads and speaks English.
  * Willing and able to provide informed consent according to institutional guidelines.

Exclusion Criteria:

* Child Participant:

  * Patients diagnosed with cancer who have relapsed or have recurrence of disease within the past month or those with progressive disease.
  * Patients in medical crisis as determined by consultation with their primary care physician.
  * On bone marrow transplant service.
  * On inpatient service or expected/scheduled inpatient admission (e.g. hospitalized).
  * Acute complications of sickle cell disease requiring hospitalization or an acute care visit including pain crises, acute chest syndrome, acute cerebrovascular events/stroke or active infection/fever.
  * Patient is residing in St. Jude long-term nonsmoking housing facility (e.g. Target House or Ronald McDonald House) during the 7-day texting data collection phase.
* Parent participant:

  * Cannot be in crisis or distress or have another disabling condition that would preclude participation as determined by review of patient's medical record prior to study enrollment.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: For the purposes of this protocol, the notation of the term "parent" will be used to include biological parents, step-parents, and legal guardians. The primary study population will consist of patients and parents with the characteristics noted under eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Rate of participation and compliance by disease group | at end of 7-day period
  Rates of participation on the study, compliance with reporting SHSe, feedback about the technical viability of the texting methods, and satisfaction regarding the texting procedures will be obtained.

SECONDARY OUTCOMES:
Parent reports of child SHSe; attitudinal, behavioral, and other socio-environmental variables. | at end of 90-day period

CONTACTS AND LOCATIONS:
Overall Officials: James Klosky, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols